CLINICAL TRIAL: NCT00731666
Title: Prospective, Non-randomized, Multi-center Clinical Trial to Assess the Effectiveness of the Coloplast Titan® IPP at Maintaining or Increasing Penile Length After Implantation
Brief Title: Evaluation of the Coloplast Titan® IPP for Maintaining Penile Length While Treating Erectile Dysfunction (ED)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: US001SU
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-09

CONDITIONS: Erectile Dysfunction
Keywords: penile length; IPP; Erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Titan® IPP (Other): Subjects implanted with Titan® IPP
  Interventions: Device: Inflatable Penile Prosthesis

INTERVENTIONS:
Device: Inflatable Penile Prosthesis — Hydraulic system designed to be surgically implanted into the penis for the management of erectile dysfunction. The implant provides the participant with voluntary control over the erect and flaccid states of the penis.
  Other Names: Titan

SUMMARY:
This study is designed to assess the effectiveness of the Coloplast Titan® Inflatable Penile Prosthesis (IPP) at maintaining or increasing penile length after implantation of the device. It will incorporate a modified method of cylinder sizing during implantation and a max-inflate technique after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Has an estimated life expectancy of more than 5 years
* Has been diagnosed with erectile dysfunction
* Is willing to have the Titan IPP implanted
* Is able and willing to complete all follow-up visits and procedures indicated in this protocol
* Has been informed of the nature of the study and agrees to its provisions and - Has provided written informed consent as approved by the Institutional Review board of the respective site

Exclusion Criteria:

* Participant has had a previous penile prosthesis or prior penile enlargement surgeries
* Participant has a compromised immune system
* Participant has had a myocardial infarction or coronary artery stent placement within 2 months prior to treatment
* Participant does not have manual dexterity or mental ability to operate the pump
* Participant has an active urogenital infection or active skin infection in region of surgery
* Participant is diagnosed with fibrotic disease, such as priapism or Peyronie's disease
* Participant is diagnosed with Chordee
* Participant has neuropathy
* Participant has a serious bleeding disorder or coagulopathy

Ages: 25 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-12; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Henry, MD, Principal Investigator — Regional Urology, LLC; Rafael Carrion, MD, Principal Investigator — JAames A Haley VA; Run Wang, MD, Principal Investigator — University of Texas
Locations (3):
- United States (3):
  - James A Haley VA, Tampa, Florida
  - Regional Urology, LLC, Shreveport, Louisiana
  - University of Texas Health Science Center at Houston, Houston, Texas

REFERENCES:
- [Derived] Henry GD, Carrion R, Jennermann C, Wang R. Prospective evaluation of postoperative penile rehabilitation: penile length/girth maintenance 1 year following Coloplast Titan inflatable penile prosthesis. J Sex Med. 2015 May;12(5):1298-304. doi: 10.1111/jsm.12833. Epub 2015 Apr 14. PMID 25872574

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Titan® IPP
Started | 40
Completed | 28
Not Completed | 12
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 8
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Titan® IPP
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 66.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: The Study's Primary Objective Will Assess the Change in Penile Length.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Titan® IPP
Number analyzed (Participants) | 31
cm
  Pubic bone to meatus - erect | 1.14 (1.94)
  Pubic bone to meatus - flaccid | 0.99 (1.64)
  Pubic bone to meatus - stretched | 1.04 (1.94)
  Pubic bone to proximal end of corona - erect | 0.94 (1.41)
  Pubic bone to proximal end of corona - flaccid | 0.69 (1.69)
  Pubic bone to proximal end of corona - stretched | 0.59 (1.59)
  Pubopenile skin junction to meatus - erect | 0.93 (1.41)
  Pubopenile skin junction to meatus - flaccid | 0.71 (1.48)
  Pubopenile skin junction to meatus - stretched | 0.95 (1.98)
  Pubopenile skin junct to prox end of corona-erect | 0.93 (1.5)
  Pubopenile skin junct to prox end of corona-flacci | 0.75 (1.58)
  Pubopenile skin junct to prox end of corona-stretc | 0.64 (2.00)

2. Secondary Outcome: Assess Participant Satisfaction With the Penile Length at Baseline, 12 and 24 Months Post Implantation Via Participant Questionaire.
Time Frame: 12 and 24 months
Population: Subjects implanted with Titan IPP
Measure: Number; unit: percentage of participants
Arm/Group | Titan® IPP
Number analyzed (Participants) | 31
percentage of participants
  At 12 mo: Over past 4 wks, completely satisfied | 48.4
  At 12 mo: Over past 4 wks, mostly satisfied | 16.1
  At 12 mo: Over past 4 weeks, somewhat dissatisfied | 22.6
  At 12 mo: Over past 4 wks, completely dissatisfied | 12.9
  At 24 mo: Over past 4 wks, completely satisfied | 57.1
  At 24 mo: Over past 4 wks, mostly satisfied | 10.7
  At 24 mo: Neutral | 3.6
  At 24 mo: Over past 4 weeks, somewhat dissatisfied | 7.1
  At 24 mo: Over past 4 weeks, completely dissatisfi | 21.4

3. Secondary Outcome: The Rate of Change in Male Stress Urinary Incontinence(SUI).
Description: Subject responses to 3 questions were evaluated:
  1. On average, how many of these (pads, tissues, disposable undergarments) would you use to protect against wetness during the day?
  2. Overall, how often have you needed to change your daily activities because of urinary incontinence?
  3. Overall, how big of a social problem has urinary incontinence been for you during the past month?
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Titan® IPP
Number analyzed (Participants) | 31
percentage of participants
  Question 1: Improved | 16.7
  Question 1: Unchanged (Satisfactory) | 66.7
  Question 1: Worsened | 16.7
  Question 2: Improved | 12.9
  Question 2: Unchanged (Satisfactory) | 61.3
  Question 2: Worsened | 25.8
  Question 3: Improved | 19.4
  Question 3: Unchanged (Satisfactory) | 67.7
  Question 3: Unchanged (Unsatisfactory) | 3.2
  Question 3: Worsened | 9.7

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 24 months.
Arm/Group | Titan® IPP
Serious Adverse Events (participants affected / at risk) | 1/40
Other Adverse Events (participants affected / at risk) | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Titan® IPP (N=40)
Infection (Surgical and medical procedures) | 1 (1) — Procedure-related infection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No